CLINICAL TRIAL: NCT00386243
Title: Evaluation of Stepped Care for Chronic Pain in Iraqi/Afghanistan Veterans
Brief Title: Evaluation of Stepped Care for Chronic Pain in Iraq/Afghanistan Veterans (ESCAPE)
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F4437-I; NCT00449475 (obsolete NCT alias)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-05

CONDITIONS: Low Back Pain; Pain; Pain, Intractable
Keywords: analgesia; analgesics; cognitive behavioral therapy; Pain; self-management; stepped care; musculoskeletal pain
MeSH Terms: conditions — Low Back Pain; Pain; Pain, Intractable; Agnosia; Musculoskeletal Pain | interventions — Cognitive Behavioral Therapy; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Study subjects randomized to this arm would receive usual care from their provider(s). No study intervention is undertaken on subjects in this arm. Participants in Usual Care would complete the same four outcome assessments (surveys) throughout the course of the study that members of the intervention complete.
- Stepped Care (Experimental): Study subjects randomized to this arm would receive stepped care for their pain. Stepped care involves FDA-approved analgesic therapy, a 12-week pain self-management program, and if pain does not improve, a 12-week cognitive behavioral therapy program.
  Interventions: Behavioral: Cognitive behavioral therapy; Behavioral: Pain self-management program; Drug: Co-Analgesic Therapy; Drug: Opioid Analgesics

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy is delivered by phone by a nurse care-manager 6 times over a 12-week period. Sessions last approximately 45 minutes and occur at weeks 14, 16, 18, 20, 22, and 24 of the study.
  Other Names: Often referred to as "CBT."
  Arms: Stepped Care
Behavioral: Pain self-management program — The pain self-management program is delivered by a nurse care-manager during a 12-week period. Sessions are each 45 minutes long and phone-based. They occur at baseline, week 1, week 3, week 6, week 9, and week 12.
  Arms: Stepped Care
Drug: Co-Analgesic Therapy — Amitriptyline, start at 10-25, titrate to 100 mg Nortriptyline, start at 10-25, titrate to 100 mg
  Gabapentin, titrate up to 900-1200 tid venlafaxine, carbemazepine, duloxetine, and/or pregabalin
  Cyclobenzaprine, titrate to 10 mg TID fluoxetine, sertraline, citalopram
  Arms: Stepped Care
Drug: Opioid Analgesics — Tramadol 50 mg BID or TID and titrate to 100 mg QID Acetaminophen/codeine (300mg/30mg). Take 1 or 2 tablets qid prn pain Acetaminophen/hydrocodone (500mg/5mg). Take 1 or 2 tablets qid prn pain Acetaminophen/oxycodone (500mg/5mg). Take 1 or 2 tablets qid prn pain Morphine SR (30mg). Start at 30 mg twice a day (titrate up to 240mg/day if needed) Methadone (5-10mg). Start at 5mg bid; titrate 10mg tid (max 20mg tid)
  Arms: Stepped Care

SUMMARY:
The purpose of this study is to determine if a stepped-care intervention makes pain symptoms better and reduces activity limitations because of pain. Our two primary hypotheses are that in OIF/OEF veterans with chronic pain:

1. Stepped care is more effective than usual care in reducing pain-related disability
2. Stepped care is more effective than usual care in reducing psychological distress

DETAILED DESCRIPTION:
Through the Evaluation of Stepped Care for Chronic Pain (ESCAPE) trial we aim to develop and test a stepped-care intervention to improve functional and work-related outcomes in Operation Iraqi Freedom/Operation Enduring Freedom veterans with chronic musculoskeletal pain. Stepped-care involves starting with lower intensity, less costly treatments initially (Step 1) and "stepping up" to more intensive, costly, or complex treatments in patients with inadequate response (Step 2). The study design will be a randomized controlled trial. The stepped care approach will involve 12 weeks of a pain self-management program in Step 1 followed by 12 weeks of brief cognitive behavioral therapy in participants with inadequate improvement in pain-related disability (Step 2). Patients treated in usual care will be the control group. Thus, the primary objective of the ESCAPE trial is to conduct a randomized controlled trial to compare the effectiveness of a stepped care intervention vs. usual care in OIF/OEF veterans with chronic and disabling musculoskeletal pain and evaluate the impact of this intervention on pain-related disability, work function, psychological distress, and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* have musculoskeletal pain of the low back, cervical spine, or extremities
* have chronic pain (>3 months duration)
* have moderate functional impairment
* have access to a working telephone
* Indianapolis Roudebush VA Medical Center patient or Walter Reed Army Medical Center patient
* willing to travel at least once to study site

Exclusion Criteria:

* prior back or cervical spine surgery or surgery pending
* active psychosis
* incompetent for interview
* severe impairment of hearing or speech
* active suicidal ideation
* current alcohol or other substance dependence or abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2007-12; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Bair, MD MS, Principal Investigator — Richard Roudebush VA Medical Center
Locations (1):
- Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Kroenke K, Bair MJ, Damush TM, Wu J, Hoke S, Sutherland J, Tu W. Optimized antidepressant therapy and pain self-management in primary care patients with depression and musculoskeletal pain: a randomized controlled trial. JAMA. 2009 May 27;301(20):2099-110. doi: 10.1001/jama.2009.723. PMID 19470987
- [Derived] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Derived] Bair MJ, Ang D, Wu J, Outcalt SD, Sargent C, Kempf C, Froman A, Schmid AA, Damush TM, Yu Z, Davis LW, Kroenke K. Evaluation of Stepped Care for Chronic Pain (ESCAPE) in Veterans of the Iraq and Afghanistan Conflicts: A Randomized Clinical Trial. JAMA Intern Med. 2015 May;175(5):682-9. doi: 10.1001/jamainternmed.2015.97. PMID 25751701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began December 2007 and concluded June 2011. The final assessment was completed by May 2012. All subjects were recruited from the Roudebush VA Medical Center.
Groups:
- Stepped Care: Study subjects randomized to this arm would receive stepped care for their pain. Stepped care involves FDA-approved analgesic therapy, a 12-week pain self-management program, and if pain does not improve, a 12-week cognitive behavioral therapy program.
  Pain self-management program : The pain self-management program is delivered by a nurse care-manager during a 12-week period. Sessions are each 45 minutes long and phone-based. They occur at baseline, week 1, week 3, week 6, week 9, and week 12.
  Cognitive behavioral therapy : Cognitive behavioral therapy is delivered by phone by a nurse care-manager 6 times over a 12-week period. Sessions last approximately 45 minutes and occur at weeks 14, 16, 18, 20, 22, and 24 of the study.
  Co-Analgesic Therapy
Period: Overall Study
Arm/Group | Usual Care | Stepped Care
Started | 121 | 121
Completed | 114 | 108
Not Completed | 7 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Stepped Care | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 120 | 241
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (10.5) | 36.4 (10.1) | 36.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 105 | 109 | 214
Region of Enrollment [Number; unit: participants]
  United States | 121 | 121 | 242

OUTCOME MEASURES:

1. Primary Outcome: Roland-Morris Disability Questionnaire
Description: This is a 24-item pain specific disability questionnaire consisting of 24 questions which are related specifically to physical functions that are likely to be affected by back pain. The questionnaire is scored by adding up the number of items checked by the subject (0-24 range). Greater levels of disability are reflected by higher numbers.
Time Frame: at baseline and 9 months
Population: We had baseline data available for 241 participants; 120 in the usual care arm and 121 in the stepped care arm. At 9 months, 7 participants withdrew from the study leaving 114 usual care participants available for analysis. In the stepped care arm, 13 participants withdrew leaving 108 available for analysis
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
scores on a scale
  baseline | 13.7 (4.7) | 14.0 (4.3)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 12.1 (6.4) | 10.6 (6.3)

2. Primary Outcome: Brief Pain Inventory (Interference)
Description: This is an 7-item measure that provides scores for pain-related functional impairment. The seven (7) pain interference items are rated on a simple numeric rating scale from 0-10. On the scale 0 represents "no interference" and 10 is "completely interferes". The pain interference score is achieved by taking the total of all seven (7) scores and dividing it by the number of items (7).
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
units on a scale
  At Baseline | 5.4 (2.4) | 5.3 (2.1)
  At 9 months: number analyzed (Participants) | 114 | 108
  At 9 months | 4.5 (2.7) | 3.8 (2.6)

3. Secondary Outcome: SF-Mental Component Summary (MCS)
Description: This scale provides a measure of mental health quality of life. It is measure on a 0 to 100 scale with higher scores representing better mental health
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
units on a scale
  Baseline | 41.4 (13.2) | 41.9 (12.1)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 42.4 (12.5) | 42.2 (13.1)

4. Secondary Outcome: PHQ-9 Depression
Description: This measure assesses depression symptoms on a 0 to 27 scale with higher scores representing more severe depression
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
scores on a scale
  Baseline | 11.3 (5.64) | 11.05 (6.18)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 10.0 (6.34) | 9.45 (6.84)

5. Secondary Outcome: PTSD Checklist-17 Civilian Version (PCL-C)
Description: The PCL-17 is a standardized self-report rating scale for PTSD comprising 17 items that correspond to the key symptoms of PTSD. Two versions of the PCL exist: PCL-Military and PCL-Civilian.We used the PCL-Civilian version because it addresses the broadest range of possible events as the traumatic stressor. The PCL-C has demonstrated strong reliability and validity in multiple samples. A total symptom severity score (range = 17-85) can be obtained by summing the scores from each of the 17 items that have response options ranging from 1 "Not at all" to 5 "Extremely". Higher scores represent more severe PTSD symptoms.
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
score on a scale
  Baseline | 25.15 (19.74) | 27.62 (19.24)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 22.71 (19.15) | 24.28 (19.07)

6. Secondary Outcome: GAD-7 Anxiety Score
Description: This 7-item scale assesses anxiety symptoms on a 0 to 21 scale with higher scores representing more severe anxiety symptoms
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
units on a scale
  Baseline | 8.66 (5.22) | 8.95 (5.30)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 7.85 (5.5) | 7.89 (5.55)

7. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0-52 with higher scores representing more pain catastrophizing.
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Stepped Care
Number analyzed (Participants) | 120 | 121
units on a scale
  Baseline | 21.81 (12.38) | 21.44 (12.26)
  9 months: number analyzed (Participants) | 114 | 108
  9 months | 18.40 (13.46) | 16.63 (12.29)

ADVERSE EVENTS:
Time Frame: The time frame in which adverse event data were collected was from the baseline evaluation to the 9-month assessment. Therefore, the assessment period was for 9 months which was through study completion.
Description: There were 7 Serious Adverse Events reported to the IRB according to the VA definition of a serious adverse event. VA requires reporting of any hospital stay longer than 24 hours by any subject enrolled. There were 7. The IRB did not find these to be Serious Adverse Events resulting from the study and these are called "VA Events" officially.
Arm/Group | Usual Care | Stepped Care
Serious Adverse Events (participants affected / at risk) | 1/121 | 6/121
Other Adverse Events (participants affected / at risk) | 0/121 | 4/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=121) | Stepped Care (N=121)
hospital stay longer than 24 hours (Psychiatric disorders) | 1 (1) | 3 (3) — IRB found that this event not to be a serious adverse event
hospitalization for longer than 24 hours (Nervous system disorders) | 0 (0) | 2 (2) — IRB found these not to be serious adverse events
hospitalization for longer than 24 hours (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — IRB concluded that this did not meet their definition for a serious adverse event
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=121) | Stepped Care (N=121)
Medication side effects (Nervous system disorders) | 0 (0) | 2 (2) — dizziness related to study medication
Medication side effects (Gastrointestinal disorders) | 0 (0) | 2 (2) — nause related to study medication

LIMITATIONS AND CAVEATS:
Single VA Center; May not generalize to non-VA samples

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No